CLINICAL TRIAL: NCT05674136
Title: Clinical Equivalence of Masimo INVSENSOR00061 to RD SET Neo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIP-1056
Record Dates: First submitted 2022-12-08; First posted 2023-01-06 (Actual); Results first posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Test Subject (Experimental): All subjects who are enrolled into the test group and participate in data collection receive the noninvasive INVSENSOR00061 sensor
  Interventions: Device: INVSENSOR00061

INTERVENTIONS:
Device: INVSENSOR00061 — Noninvasive pulse oximeter sensor

SUMMARY:
This study is designed to compare the equivalence of the Masimo INVSENSOR00061 to RD SET Neo for SpO2 and performance of PR and RRp as the subjects undergo a controlled desaturation protocol. This type of study design is required to evaluate the performance of pulse oximeters based upon the ISO 80601-2-61 standard which is also adopted and referenced by the FDA.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 to 50 years of age.
* Subject weighs a minimum of 110 lbs.
* Hemoglobin value ≥ 11 g/dL.
* Baseline heart rate ≥ 45 bpm and ≤ 85 bpm.
* Blood Pressure: Systolic BP ≤ 140 mmHg and ≥ 90 mmHg, Diastolic BP ≤ 90 mmHg and ≥ 50 mmHg, and if systolic BP is lower than 100 mmHg and/or diastolic BP is lower than 60 mmHg, subject passes an orthostatic blood pressure test.
* CO value ≤ 3.0% FCOHb.
* Subject is able to read and communicate in English and understands the study and the risks involved

Exclusion Criteria:

* Subject is pregnant.
* Subject has a BMI > 35.
* Subject is wearing nail polish that cannot be removed, gel nails, and/or acrylic nails that can interfere with study device's placement is deemed ineligible at the discretion of investigator/study staff. *
* Subject has a history of fainting (vasovagal syncope), blacking out or losing consciousness during or after a blood draw, or has a fear of blood draws.
* Subject has open wounds, inflamed tattoos or piercings, and/or has any visible healing wounds that a medical professional determines may place them at an increased risk for participation. *
* Subject has known drug or alcohol abuse.
* Subject uses recreational drugs. *
* Subject experiences frequent or severe headaches and/or migraine headaches, migraine auras, altitude sickness, and/or headaches accompanied by visual changes or sensitivity to light or sound.
* Subject has experienced a concussion or head injury with loss of consciousness within the past 12 months.
* Subject has any history of a stroke, myocardial infarction (heart attack), and/or seizures.
* Subject has any chronic bleeding disorder (e.g., hemophilia).
* Subject has taken anticoagulant medication within the past 30 days (excluding nonsteroidal anti-inflammatory drugs (NSAIDS)).
* Subject has donated blood within the past 4 weeks.
* Subject has Wolff-Parkinson-White Syndrome or Stokes-Adams Syndrome.
* Subject has any cardiac dysrhythmia (e.g., atrial fibrillation) and has not received clearance from their physician to participate.
* Subject has a known neurological and/or psychiatric disorder (e.g., schizophrenia, bipolar disorder, Multiple Sclerosis, Huntington's disease) that interferes with the subject's level of consciousness. *
* Subject has taken opioid pain medication 24 hours before the study.
* Subject has any active signs and/or symptoms of infectious disease (e.g., Hepatitis, HIV, Tuberculosis, Flu, Malaria, Measles, etc.). *
* Subject is taking medications known to treat any type of infectious disease.
* Subject has either signs or history of peripheral ischemia or carpal tunnel syndrome.
* Subject has had invasive surgery within the past year, including but not limited to major dental surgery, appendectomy, plastic surgery, jaw surgery, major ENT surgery, major abdominal and/or pelvic surgery, heart surgery, or thoracic surgery. *
* Subject has symptoms of congestion, head cold, or other illnesses.
* Subject has been in a severe car accident(s) or a similar type of accident(s) requiring hospitalization within the past 12 months.
* Subject has any cancer or history of cancer (not including skin cancer). *
* Subject has chronic unresolved asthma, lung disease (including COPD) and/or respiratory disease.
* Subject is allergic to lidocaine, chlorhexidine, latex, adhesives, or plastic.
* Subject has a heart condition, insulin-dependent diabetes, or uncontrolled hypertension.
* Subject has delivered vaginally, has had a pregnancy terminated, a miscarriage with hospitalization or had a C-section within the past 6 months.
* Subject intends on participating in any heavy lifting, repetitive movement of their wrist (including riding a motorcycle, tennis), exercise (working out, riding a bike, riding a skateboard, etc.), or any activity that will put additional stress on the wrist within 24 hours following a study that involves an arterial line.
* Subject has any medical condition which in the judgment of the investigator and/or medical staff, renders them ineligible for participation in this study or subject is deemed ineligible by the discretion of the investigator/study staff.

(*)Physician's discretion.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2022-11-18 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Masimo Corporation, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Masimo INVSENSOR00061: All subjects who are enrolled into the test group and participate in data collection receive the noninvasive Masimo INVSENSOR00061 sensor
  Masimo INVSENSOR00061: Noninvasive pulse oximeter sensor
Period: Overall Study
Arm/Group | Masimo INVSENSOR00061
Started | 62
Completed | 42
Not Completed | 20

BASELINE CHARACTERISTICS:
Population: 3 subjects not used for baseline analysis due to sensor placement issues. 9 subjects not used for baseline analysis due to incorrect software version.
Arm/Group | Masimo INVSENSOR00061
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 7
  More than one race | 2
  Unknown or Not Reported | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: SpO2 Accuracy
Description: SpO2 accuracy was determined by calculating the root mean-squared (rms) difference between the measured values (SpO2i) to the reference values (SpO2ref_i) in accordance with ISO-80601-2-61. Arms= √(∑(i=1 to n) ((SpO2_i-SpO2ref_i )^2 ))/n
Time Frame: 1-3 hours
Measure: Number; unit: % of oxygen saturated hemoglobin
Arm/Group | Test Subject
Number analyzed (Participants) | 30
% of oxygen saturated hemoglobin | 1.24

ADVERSE EVENTS:
Time Frame: 1-3 hours
Arm/Group | Masimo INVSENSOR00061
All-Cause Mortality (participants affected / at risk) | 0/62
Serious Adverse Events (participants affected / at risk) | 0/62
Other Adverse Events (participants affected / at risk) | 6/62
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Masimo INVSENSOR00061 (N=62)
Venipuncture or Intravenous puncture (Injury, poisoning and procedural complications) | 4
Lightheadedness (Injury, poisoning and procedural complications) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-04): https://cdn.clinicaltrials.gov/large-docs/36/NCT05674136/Prot_SAP_000.pdf